CLINICAL TRIAL: NCT04216641
Title: Impact of a Food Improvement Strategy on Their Appreciation in a Population of Cancer Patients Treated With Chemotherapy
Brief Title: Cancer, Nutrition and Taste
Acronym: CANUT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL19_0292
Record Dates: First submitted 2019-10-01; First posted 2020-01-03 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Cancer; Nutrition Disorders
Keywords: cancer, nutrition disorder
MeSH Terms: conditions — Neoplasms; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): At each meal: different elements will be presented to the patient (starter / main course / side dish / dessert).
  For each of these elements, the patient will be offered 4 versions (a standard version and 3 adapted versions of the same food):
  * The standard food.
  * The food refers to a more elaborate texture.
  * The food refers to a food with a stronger smell.
  * The food refers to a more important flavor.
  The patient will indicate the version of the food that will be preferred.
  Interventions: Dietary Supplement: Adapted food intervention

INTERVENTIONS:
Dietary Supplement: Adapted food intervention — Adapted food intervention

SUMMARY:
Cancer promotes weight loss; it can also lead to particular complications for patients during treatment. A team led by Dr Michael Sawyer, showed the deleterious impact of undernutrition on the benefits of chemotherapy.

Cancer patients are at high risk of undernutrition, which is generally more pronounced for solid tumours (upper digestive tract, ENT, bronchial tubes…). This undernutrition leads to major weight loss and wasting, and may represent the first sign of a call for a diagnosis of cancer. Cancer-related undernutrition is multi-factorial in origin and has multiple consequences; it has its own prognostic value.

Chemotherapy treatments can induce various adverse effects in patients, including sensory disturbances at the beginning of treatment in addition to disturbances that may already be present before any treatment. Altered taste and odour, observed in 86% of patients, can induce a change in food preferences, promote the development of aversions, and therefore, lead to a significant reduction in the pleasure of eating. Loss of appetite, decreased food intake and the development of aversions to certain foods are situations experienced by a large proportion of patients undergoing chemotherapy.

The assessment of taste disorders in patients undergoing chemotherapy treatment is established through the use of questionnaires, interviews and taste tests.

Changes in the perception and identification of salty, sweet, bitter and sour flavours are common in patients undergoing chemotherapy.

The objective of CANUT is to study the effect of pathology and chemotherapy on gustatory and olfactory mechanisms and in particular on interindividual differences in the perception and appreciation of food.

In this study the investigators propose to adapt foods to best respond to sensory disorders related to the disease and/or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with advanced lung cancer requiring a first line of intravenous chemotherapy or patient with localized, histologically or cytologically proven breast cancer for whom intravenous chemotherapy treatment will be initiated or patient with stage III-IV gynecological cancer (ovarian cancer or uterine cancer) for whom intravenous chemotherapy treatment will be initiated.

  * Patient with a body mass index (BMI) between 18Kg/m² and 35Kg/m².
  * Patient whose indication for treatment with intravenous chemotherapy has been selected
  * Naive patient of previous chemotherapy.
  * Life expectancy > 3 months.
  * Patient able to travel for 4 visits to the Paul Bocuse Institute, 1 Chemin de Calabert, 69 130 ECULLY, FRANCE.
  * Written informed consent obtained in accordance with applicable GCPs.
  * Patients affiliated to a social security system.
  * Patients who have the possibility of being accompanied, by the same person, to the visits of the test meals at the Paul Bocuse Research Institute

Exclusion Criteria:

* Patient under 18 years of age.
* Patient who has had another malignant tumor in the last 3 years.
* Patient with symptomatic brain metastases.
* Patient with symptomatic mucositis.
* Patient suffering or having suffered from an otorhinolaryngic or oesogastrointestinal pathology interfering with food intake.
* Patients with digestive disorders before any cancer treatment.
* Indication for concomitant radiotherapy or immunotherapy alone treatment.
* Patient with a known food allergy or food intolerance.
* Patient with partial or total agueusia diagnosed.
* Patient with diagnosed partial or total anosmia.
* Patients who have used artificial feeding within 2 months.
* Patients who have lost more than 10% of their baseline weight within 2 months.
* Patient unable to be regularly monitored for any reason
* Patient deprived of liberty or placed under guardianship or curatorship
* Pregnant or breastfeeding patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
proportion of treated patients by 4 cycles of chimiotherapy that will prefere at least 1 modified version of meal. | 12 weeks
  The main endpoint of the CANUT-1 study is the proportion of cancer patients treated with chemotherapy (after 4 cycles) who will prefer at least an adapted version of a food compared to the standard version of the same food.

SECONDARY OUTCOMES:
Food assessment scores ( 0/4 to 4/4, 4 mean a better score) | Before Cycle 1(each cycle is 28 days) of chemotherapy treatment
  Individual food assessment scores (standard food and adapted food to taste and smell disorders) before any treatment
Food assessment scores ( 0/4 to 4/4,4 mean a better score) | after 2 cycles (each cycle is 28 days) of chemotherapy
  : Individual food assessment scores (standard food and adapted food to taste and smell disorders) after 2 cycles of chemotherapy
Food assessment scores ( 0/4 to 4/4, 4 mean a better score) | after 4 cycles(each cycle is 28 days) of chemotherapy
  : Individual food assessment scores (standard food and adapted food to taste and smell disorders) after 4 cycles of chemotherapy
European Test of Olfactory Capabilities (ETOC) (1 (mean a worse) to 9 (mean a better) | Before cycle 1(each cycle is 28 days) of chemotherapy treatment
  The results of olfactory detection and identification, familiarity, pleasantness, intensity, edibility and trigeminal perception (fresh, hot, irritant, pungent) European Test of Olfactory Capabilities (ETOC) before any treatment, after 2 and 4 cycles of chemotherapy.
  The results of olfactory detection and identification, familiarity, pleasantness, intensity, edibility and trigeminal perception (fresh, hot, irritant, pungent) European Test of Olfactory Capabilities (ETOC) before any treatment
European Test of Olfactory Capabilities (ETOC)(1 (mean a worse) to 9 (mean a better) | after 2 cycles (each cycle is 28 days) of chemotherapy
  The results of olfactory detection and identification, familiarity, pleasantness, intensity, edibility and trigeminal perception (fresh, hot, irritant, pungent) European Test of Olfactory Capabilities (ETOC) after 2 of chemotherapy.
European Test of Olfactory Capabilities (ETOC)(1 (mean a worse) to 9 (mean a better) | after 4 cycles(each cycle is 28 days) of chemotherapy
  The results of olfactory detection and identification, familiarity, pleasantness, intensity, edibility and trigeminal perception (fresh, hot, irritant, pungent) European Test of Olfactory Capabilities (ETOC) after and 4 cycles of chemotherapy.
Condiments consumption assessment by condiments questionnaire (0 contiment to 12 condiments) | Before cycle 1(each cycle is 28 days) of treatment
  The number of condiments added at the time of inclusion
Condiments consumption assessment by condiments questionnaire (0 contiment to 12 condiments) | after 2 cycles(each cycle is 28 days) of chemotherapy
  The number of condiments added after 2 cycles of chemotherapy.
Condiments consumption assessment by condiments questionnaire (0 contiment to 12 condiments) | after 4 cycles(each cycle is 28 days) of chemotherapy
  The number of condiments added after 4 cycles of chemotherapy.
Food temperature | Before Cycle 1(each cycle is 28 days) of chemotherapy treatment
  The proportion of patients who prefer to consume cold foods versus those who prefer to consume hot foods at the time of inclusion
Food temperature | after 2 cycles(each cycle is 28 days) of chemotherapy
  The proportion of patients who prefer to consume cold foods versus those who prefer to consume hot foods after 2 cycles of chemotherapy
Food temperature | after 4 cycles(each cycle is 28 days) of chemotherapy
  The proportion of patients who prefer to consume cold foods versus those who prefer to consume hot foods at 4 cycles of chemotherapy

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Louis Pradel, Bron
  - Hôpital de jour - Hôpital de la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon

IPD SHARING:
Plan to Share IPD: No